CLINICAL TRIAL: NCT04684485
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of SCD-044 in the Treatment of Moderate to Severe Atopic Dermatitis
Brief Title: To Assess the Efficacy and Safety of SCD-044 in the Treatment of Moderate to Severe Atopic Dermatitis
Acronym: SOLARES-AD-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCD-044-19-16
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo of SCD-044 product (Placebo Comparator): Placebo tablet of SCD-044 product in subjects with moderate to severe atopic dermatitis.
  Interventions: Drug: Placebo
- SCD-044 Tablets_Dose 1 (Active Comparator): SCD-044 Tablets of low dose (Dose 1) in subjects with moderate to severe atopic dermatitis.
  Interventions: Drug: SCD-044_Dose 1
- SCD-044 Tablets_Dose 2 (Active Comparator): SCD-044 Tablets of intermediate dose (Dose 2) in subjects with moderate to severe atopic dermatitis.
  Interventions: Drug: SCD-044_Dose 2
- SCD-044 Tablets_Dose 3 (Active Comparator): SCD-044 Tablets of high dose (Dose 3) in subjects with moderate to severe atopic dermatitis.
  Interventions: Drug: SCD-044_Dose 3

INTERVENTIONS:
Drug: Placebo — Placebo Tablet of SCD-044 product in subjects with moderate to severe atopic dermatitis.
  Arms: Placebo of SCD-044 product
Drug: SCD-044_Dose 1 — SCD-044 tablets of low dose (Dose 1) in subjects with moderate to severe atopic dermatitis.
  Arms: SCD-044 Tablets_Dose 1
Drug: SCD-044_Dose 2 — SCD-044 tablets of intermediate dose (Dose 2) in subjects with moderate to severe atopic dermatitis.
  Arms: SCD-044 Tablets_Dose 2
Drug: SCD-044_Dose 3 — SCD-044 tablets of high dose (Dose 3) in subjects with moderate to severe atopic dermatitis.
  Arms: SCD-044 Tablets_Dose 3

SUMMARY:
This is a Phase II, randomized, double-blind, placebo-controlled study in subjects with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
This is a Phase II, randomized, double-blind, placebo-controlled study to determine the effect of SCD-044 in subjects with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 18 years.
2. Males and non-pregnant non-lactating females, diagnosed with chronic atopic dermatitis for ≥ 1 year at Screening and Baseline based on Eichenfield revised criteria of Hanifin and Rajka.
3. Moderate to severe atopic dermatitis at Screening and Baseline

Exclusion Criteria:

1. Female Subjects who are pregnant, nursing, or planning to become pregnant during study participation or within 6 months of completing the study.
2. Known organ complications of Diabetes mellitus such as reduced renal function, significant retinal pathology or neuropathy.
3. History or presence of uveitis

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2025-03-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (58):
- United States (34):
  - Omni Dermatology, Phoenix, Arizona
  - Yuma Clinical Trials, LLC, Yuma, Arizona
  - T. Joseph Raoof Md, Imc./Encino Research Center, Encino, California
  - Metropolis Dermatology, Los Angeles, California
  - Axis Clinical Trials, Los Angeles, California
  - Providence Clinical Research, North Hollywood, California
  - Unison Clinical Trials, Sherman Oaks, California
  - Providere' Research Inc., West Covina, California
  - Clarity Dermatology, Castle Rock, Colorado
  - Accel Research Sites Network - Annexus Dermatology & Aestheitcs, DeLand, Florida
  - Revival Research Corporation, Doral, Florida
  - Advanced Clinical Research Institute, Florida City, Florida
  - FXM Clinical Research Fort Lauderdale, Fort Lauderdale, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Evolution Research Center, Hialeah, Florida
  - Sweet Hope Research Specialty, Inc, d/b/a Neoclinical Research, Hialeah, Florida
  - Evolution Clinical Trials, Inc, Hialeah Gardens, Florida
  - Advanced Clinical Research Network, Corp, Miami, Florida
  - MedOne Clinical Research, LLC, Miami, Florida
  - Century Research LLC, Miami, Florida
  - FXM Clinical Research Miami, Miami, Florida
  - JD Medical Group, LLC, Miami, Florida
  - FXM Clinical Research Miramar, Miramar, Florida
  - Adtremed Inc, Tampa, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - Oracle Clinical Research, College Park, Georgia
  - Physicians Research Group, West Lafayette, Indiana
  - Revival research Institute, LLC, Troy, Michigan
  - DFW Clinical Research, Dallas, Texas
  - 3A Research, El Paso, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Stride Clinical Research, Sugar Land, Texas
  - Springville Dermatology/ CCT Research, Springville, Utah
  - Skin DC Derm, Arlington, Virginia
- El Salvador (3):
  - Clinica Vargas, San Salvador
  - Clinica Dermatologica, San Salvador
  - Clinica de Dermatologia y Cirugia de Piel, Santa Tecla
- Clinical Research Centre OU, Tartu, Estonia
- Georgia (7):
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center LLC, Tbilisi
  - Israeli - Georgian Medical Research Clinic Healthycore LLC, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic LLC, Tbilisi
  - Emergency Cardiology Center by Academician G. Chapidze LLC, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - TIM - Tbilisi Institute of Medicine LLC, Tbilisi
  - David Abuladze Georgian-Italian Clinic LLC, Tbilisi
- Poland (13):
  - KLIMED, Bialystok
  - Synexus Polska Sp. z o.o. Branch in Gdansk, Gdansk
  - Dobry Lekarz' Modern Therapies Center Limited Liability Company, Krakow
  - Landa Specialist Doctor's Offices, Krakow
  - GLOBE Clinical Research, Kłodzko
  - Appletreeclinics Clinical Research Centre, Lodz
  - Dermedic Iwona Zdybska, Lublin
  - EMC Medical Institute Joint Stock Company, "Certus" Private Healthcare Facility Hospital No. 1, Poznan
  - TWOJA PRZYCHODNIA Medical Centre of Szczecin, Twoja Przychodnia SCM, Szczecin
  - National Medical Institute of the MSWiA, Clinical Department of Dermatology, Warsaw
  - Synexus Polska Sp. z o.o. Branch in Warsaw, Warsaw
  - Military Institute of Medicine - National Research Institute, Department of Dermatology CWBK, Warsaw
  - Synexus Polska Sp. z o.o. Branch in Wroclaw, Wroclaw

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1- Placebo of SCD-044 Product: Placebo tablet of SCD-044 product in subjects with moderate to severe atopic dermatitis.
  Placebo:Placebo Tabletof SCD-044product in subjects with moderate to severe atopic dermatitis
- Part 1 - SCD-044 Tablets of Low Dose (Dose 1): SCD-044 Tablets of low dose (Dose 1) in subjects with moderate to severe atopic dermatitis.
  SCD-044_Dose 1: SCD-044 tablets of low dose (Dose 1) in subjects with moderate to severe atopic dermatitis.
- Part 1 - SCD-044 Tablets of Intermediate Dose (Dose 2): SCD-044 Tablets of intermediate dose (Dose 2) in subjects with moderate to severe atopic dermatitis.
  SCD-044_Dose 2: SCD-044 tablets of intermediate dose (Dose 2) in subjects with moderate to severe atopic dermatitis.
- Part 1- SCD-044 Tablets of High Dose (Dose 3): SCD-044 Tablets of high dose (Dose 3) in subjects with moderate to severe atopic dermatitis.
  SCD-044_Dose 3: SCD-044 tablets of high dose (Dose 3) in subjects with moderate to severe atopic dermatitis.
- Part 2- Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2): Subjects initially randomized to Placebo re-randomized to SCD-044 Tablets of Intermediate Dose (Dose 2) at week16
- Part 2- Placebo to SCD-044 Tablets of High Dose (Dose 3): Subjects initially randomized to Placebo re-randomized to SCD-044 tablets of high dose(Dose 3) at week 16
- Part 2- SCD-044 Tablets of Low Dose (Dose 1): SCD-044 Tablets of low dose (Dose 1) in subjects with moderate to severe atopic dermatitis.
- Part 2- SCD-044 Tablets of Intermediate Dose (Dose 2): SCD-044 Tablets of intermediatedose (Dose 2) in subjects with moderate to severe atopicdermatitis
- Part 2- SCD-044 Tablets of High Dose (Dose 3): SCD-044 Tablets of high dose (Dose 3) in subjects with moderate to severe atopic dermatitis.
Period: Part 1
Arm/Group | Part 1- Placebo of SCD-044 Product | Part 1 - SCD-044 Tablets of Low Dose (Dose 1) | Part 1 - SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 1- SCD-044 Tablets of High Dose (Dose 3) | Part 2- Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 2- Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part 2- SCD-044 Tablets of Low Dose (Dose 1) | Part 2- SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 2- SCD-044 Tablets of High Dose (Dose 3)
Started | 61 | 72 | 64 | 53 | 0 | 0 | 0 | 0 | 0
Completed | 51 | 58 | 51 | 47 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 14 | 13 | 6 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1- Placebo of SCD-044 Product | Part 1 - SCD-044 Tablets of Low Dose (Dose 1) | Part 1 - SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 1- SCD-044 Tablets of High Dose (Dose 3) | Part 2- Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 2- Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part 2- SCD-044 Tablets of Low Dose (Dose 1) | Part 2- SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 2- SCD-044 Tablets of High Dose (Dose 3)
Started | 0 | 0 | 0 | 0 | 25 | 26 | 58 | 49 | 45
Completed | 0 | 0 | 0 | 0 | 18 | 23 | 48 | 40 | 43
Not Completed | 0 | 0 | 0 | 0 | 7 | 3 | 10 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- SCD-044 Tablets of Low Dose (Dose 1): SCD-044 Tablets of low dose (Dose 1) in subjects with moderate to severe atopic dermatitis.
  SCD-044_Dose 1: SCD-044 tablets of low dose (Dose 1) in subjects with moderate to severe atopic dermatitis.
- SCD-044 Tablets of Intermediate Dose (Dose 2): SCD-044 Tablets of intermediate dose (Dose 2) in subjects with moderate to severe atopic dermatitis.
  SCD-044_Dose 2: SCD-044 tablets of intermediate dose (Dose 2) in subjects with moderate to severe atopic dermatitis.
- SCD-044 Tablets of High Dose (Dose 3): SCD-044 Tablets of high dose (Dose 3) in subjects with moderate to severe atopic dermatitis.
  SCD-044_Dose 3: SCD-044 tablets of high dose (Dose 3) in subjects with moderate to severe atopic dermatitis.
- Total: Total of all reporting groups
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3) | Total
Number analyzed (Participants) | 61 | 72 | 64 | 53 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (15.61) | 39.5 (12.42) | 40.4 (15.10) | 39.5 (13.84) | 40.6 (14.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 48 | 40 | 35 | 162
  Male | 22 | 24 | 24 | 18 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 36 | 35 | 35 | 148
  Not Hispanic or Latino | 19 | 36 | 29 | 18 | 102
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 2 | 2 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 4 | 4 | 8 | 22
  White | 50 | 59 | 52 | 38 | 199
  More than one race | 3 | 6 | 4 | 3 | 16
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Achieve ≥75% Overall Improvement in Eczema Area and Severity Index (EASI) Score From Baseline to Week 16.
Description: Based on gross morphological findings, scores will be assigned on a 4-point scale ['0' (absent), '1' (mild), '2' (moderate) and '3' (severe)] for each clinical sign.
  The information presented represents the percentage of subjects, calculated as the proportion of subjects multiplied by 100.
Time Frame: Week16
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 61 | 72 | 64 | 53
percentage of subjects | 9.8 | 18.1 | 12.5 | 15.1
Statistical Analysis 1: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets of Low Dose (Dose 1); Test type: Superiority; p = 0.1966, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets of Intermediate Dose (Dose 2); Test type: Superiority; p = 0.5438, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets of High Dose (Dose 3); Test type: Superiority; p = 0.3713, Cochran-Mantel-Haenszel

2. Secondary Outcome: Proportion of Subjects Who Achieve Score of '0' (Clear) or '1' (Almost Clear) on a 5-point, vIGA Scale and ≥2 Point Reduction From Baseline to Week 16.
Description: Based on morphological findings (overall appearance of the lesions at a given time point), scores will be assigned on a 5-point scale ('0' [clear] to 4 [severe]).
  The information presented represents the percentage of subjects, calculated as the proportion of subjects multiplied by 100.
Time Frame: Week 16
Measure: Number; unit: percentage of subject
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 61 | 72 | 64 | 53
percentage of subject | 6.6 | 9.7 | 12.5 | 9.4
Statistical Analysis 1: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets of Low Dose (Dose 1); Test type: Superiority; p = 0.4564, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets of Intermediate Dose (Dose 2); Test type: Superiority; p = 0.2515, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets of High Dose (Dose 3); Test type: Superiority; p = 0.5055, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percent Change in Mean Eczema Area and Severity Index (EASI) Score
Description: Based on gross morphological findings, scores will be assigned on a 4-point scale ['0' (absent), '1' (mild), '2' (moderate) and '3' (severe)] for each clinical sign.
Time Frame: Week 32
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2): Subjects initially randomized to Placebo re-randomized to SCD-044 Tablets of Intermediate Dose (Dose 2) at week 16
- Placebo to SCD-044 Tablets of High Dose (Dose 3): Subjects initially randomized to Placebo re-randomized to SCD-044 tablets of high dose (Dose 3) at week 16
Arm/Group | Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Placebo to SCD-044 Tablets of High Dose (Dose 3) | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 18 | 23 | 48 | 40 | 43
Percent change | -16.61 (68.985) | 6.78 (199.014) | -64.77 (26.289) | -67.04 (23.679) | -54.40 (44.901)

4. Secondary Outcome: Proportion of Subjects Who Achieve Score of '0' (Clear) or '1' (Almost Clear) on a 5-point, Validated Investigator's Global Assessment (vlGA) Scale and ≥2 Point Reduction From Baseline.
Description: as for outcome 2
Time Frame: Week 32
Measure: Number; unit: percentage of subject
Arm/Group | Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Placebo to SCD-044 Tablets of High Dose (Dose 3) | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 18 | 23 | 48 | 40 | 43
percentage of subject | 11.1 | 4.3 | 20.8 | 27.5 | 25.6

5. Secondary Outcome: Proportion of Subjects Who Achieve ≥4-point Improvement in Peak Pruritus Numeric Rating Scale (PP-NRS) From Baseline.
Description: The information presented represents the percentage of subjects, calculated as the proportion of subjects multiplied by 100.
Time Frame: Week 32
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Placebo to SCD-044 Tablets of High Dose (Dose 3) | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 16 | 22 | 45 | 38 | 42
percentage of subjects | 6.3 | 4.5 | 55.6 | 57.9 | 50.0

6. Secondary Outcome: Proportion of Subjects Who Achieve SCORing Atopic Dermatitis (SCORAD) 50 and SCORAD 75 Response at Week 32
Description: as for outcome 5
Time Frame: Week 32
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Placebo to SCD-044 Tablets of High Dose (Dose 3) | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 18 | 23 | 47 | 40 | 42
percentage of subjects
  SCORAD 50 | 16.7 | 17.4 | 51.1 | 47.5 | 50.0
  SCORAD 75 | 5.6 | 4.3 | 8.5 | 17.5 | 16.7

7. Secondary Outcome: Change From Baseline in Quality of Life Measured by Dermatology Life Quality Index (DLQI) Scores.
Description: Based on 10-item questionnaire on skin problems (0 to 3 scale). The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  The scoring of each question is as follows:
  3=Very much; 2= A lot;
  1= A little; 0= Not at all
Time Frame: Week 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Placebo to SCD-044 Tablets of High Dose (Dose 3) | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 18 | 23 | 47 | 40 | 42
score on a scale | -3.9 (4.23) | -2.2 (3.18) | -6.7 (5.93) | -6.5 (7.49) | -7.3 (6.22)

8. Secondary Outcome: Percent Change From Baseline in Body Surface Area (BSA) With Atopic Dermatitis
Time Frame: Week 32
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Placebo to SCD-044 Tablets of High Dose (Dose 3) | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 18 | 23 | 48 | 40 | 43
percent change | -19.56 (21.288) | -6.61 (95.403) | -50.14 (33.095) | -53.61 (25.314) | -43.97 (51.922)

9. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) Score
Description: Subjects will be asked to complete a 7-item questionnaire about their atopic dermatitis over the past week. Each of the seven questions carries equal weight and is scored from 0 to 4 as follows
  4= Every day; 3= 5-6 days; 2= 3-4 days;
  1= 1-2 days; 0= No days
  The POEM scores can be understood as follows:
  0 to 2= Clear or almost clear 3 to 7= Mild eczema 8 to 16= Moderate eczema 17 to 24= Severe eczema 25 to 28= Very severe eczema
  The higher the score, the more quality of life is impaired.
Time Frame: Week 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Placebo to SCD-044 Tablets of High Dose (Dose 3) | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 18 | 23 | 48 | 40 | 42
score on a scale | -2.1 (7.22) | -1.3 (3.22) | -8.4 (6.23) | -8.8 (5.93) | -8.4 (6.00)

10. Secondary Outcome: Proportion of Subjects With Improvement in Patient Global Impression of Change (PGIC) Score
Description: The subjects will be asked to assess if there has been an improvement or decline in clinical status using a 5-point scale depicting a subject's rating of overall improvement.
  The information presented represents the percentage of subjects, calculated as the proportion of subjects multiplied by 100.
Time Frame: Week 32
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Placebo to SCD-044 Tablets of High Dose (Dose 3) | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 18 | 23 | 48 | 40 | 43
percentage of participants | 88.9 | 95.7 | 85.4 | 90.0 | 88.4

11. Secondary Outcome: Patient Global Impression of Severity (PGIS) of Disease Score
Description: The subjects will be asked to assess their overall impression of disease severity over the past week using a scale of None, Mild, Moderate or Severe.
Time Frame: Week 32
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Placebo to SCD-044 Tablets of High Dose (Dose 3) | SCD-044 Tablets of Low Dose (Dose 1) | SCD-044 Tablets of Intermediate Dose (Dose 2) | SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 18 | 23 | 48 | 40 | 43
Participants
  None | 1 | 2 | 3 | 5 | 5
  Mild | 7 | 13 | 25 | 18 | 22
  Moderate | 9 | 8 | 16 | 12 | 11
  Severe | 1 | 0 | 4 | 5 | 5

12. Secondary Outcome: Adverse Events.
Description: Total Number Affected by adverse events from Baseline through Week 36
Time Frame: Week 36
Measure: Count of Participants; unit: Participants
Groups:
- Part 1-Placebo of SCD-044 Product: Placebo tablet of SCD-044 product in subjects with moderate to severe atopic dermatitis
- Part 1- SCD-044 Tablets of Low Dose (Dose 1); Part 2- SCD-044 Tablets of Low Dose (Dose 1): SCD-044 Tablets of low dose (Dose 1) in subjects with moderate to severe atopic dermatitis.
- Part 1- SCD-044 Tablets of Intermediate Dose (Dose 2); Part 2- SCD-044 Tablets of Intermediate Dose (Dose 2): SCD-044 Tablets of intermediate dose (Dose 2) in subjects with moderate to severe atopic dermatitis.
- Part 1- SCD-044 Tablets of High Dose (Dose 3); Part 2- SCD-044 Tablets of High Dose (Dose 3): SCD-044 Tablets of high dose (Dose 3) in subjects with moderate to severe atopic dermatitis.
- Part 2 - Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2): Subjects initially randomized to Placebo re-randomized to SCD-044 Tablets of Intermediate Dose (Dose 2) at week 16
- Part 2- Placebo to SCD-044 Tablets of High Dose (Dose 3): Subjects initially randomized to Placebo re-randomized to SCD-044 tablets of high dose (Dose 3) at week 16
Arm/Group | Part 1-Placebo of SCD-044 Product | Part 1- SCD-044 Tablets of Low Dose (Dose 1) | Part 1- SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 1- SCD-044 Tablets of High Dose (Dose 3) | Part 2 - Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 2- Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part 2- SCD-044 Tablets of Low Dose (Dose 1) | Part 2- SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 2- SCD-044 Tablets of High Dose (Dose 3)
Number analyzed (Participants) | 61 | 72 | 64 | 53 | 25 | 26 | 58 | 49 | 45
Participants
  Subjects with any TEAE | 13 | 23 | 18 | 18 | 4 | 5 | 13 | 17 | 11
  Subjects with serious TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 36 Weeks
Groups:
- Part 2 - Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2): Subjects initially randomized to Placebo re-randomized to SCD-044 Tablets Dose 2 (Intermediate Dose) at week 16
Arm/Group | Part 1-Placebo of SCD-044 Product | Part 1- SCD-044 Tablets of Low Dose (Dose 1) | Part 1- SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 1- SCD-044 Tablets of High Dose (Dose 3) | Part 2 - Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 2- Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part 2- SCD-044 Tablets of Low Dose (Dose 1) | Part 2- SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 2- SCD-044 Tablets of High Dose (Dose 3)
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/72 | 0/64 | 0/53 | 0/25 | 0/26 | 0/58 | 0/49 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/72 | 0/64 | 0/53 | 0/25 | 0/26 | 1/58 | 1/49 | 0/45
Other Adverse Events (participants affected / at risk) | 13/61 | 23/72 | 18/64 | 18/53 | 4/25 | 5/26 | 13/58 | 17/49 | 11/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1-Placebo of SCD-044 Product (N=61) | Part 1- SCD-044 Tablets of Low Dose (Dose 1) (N=72) | Part 1- SCD-044 Tablets of Intermediate Dose (Dose 2) (N=64) | Part 1- SCD-044 Tablets of High Dose (Dose 3) (N=53) | Part 2 - Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) (N=25) | Part 2- Placebo to SCD-044 Tablets of High Dose (Dose 3) (N=26) | Part 2- SCD-044 Tablets of Low Dose (Dose 1) (N=58) | Part 2- SCD-044 Tablets of Intermediate Dose (Dose 2) (N=49) | Part 2- SCD-044 Tablets of High Dose (Dose 3) (N=45)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1-Placebo of SCD-044 Product (N=61) | Part 1- SCD-044 Tablets of Low Dose (Dose 1) (N=72) | Part 1- SCD-044 Tablets of Intermediate Dose (Dose 2) (N=64) | Part 1- SCD-044 Tablets of High Dose (Dose 3) (N=53) | Part 2 - Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) (N=25) | Part 2- Placebo to SCD-044 Tablets of High Dose (Dose 3) (N=26) | Part 2- SCD-044 Tablets of Low Dose (Dose 1) (N=58) | Part 2- SCD-044 Tablets of Intermediate Dose (Dose 2) (N=49) | Part 2- SCD-044 Tablets of High Dose (Dose 3) (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual field defect (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis allergic (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4 | 1 | 2 | 1 | 1 | 5 | 1 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 3 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eosinophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipids increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insulin resistance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 7 | 2 | 3 | 0 | 1 | 5 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract inflammation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT04684485/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT04684485/SAP_001.pdf